CLINICAL TRIAL: NCT02001324
Title: Patient-based Outcomes for Heavy Menstrual Bleeding: Comparisons of Treatments and Methods of Data Collection
Brief Title: HMB- Data Collection Methods
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: this pilot project is no longer funded
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Kristen Matteson , M.D., Assistant Professor of Obstetrics and Gynecology, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-0062
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Heavy Menstrual Bleeding
Keywords: quality of life; heavy menstrual bleeding; electronic data collection
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paper-based data collection (Active Comparator): Paper-based data collection
  Interventions: Other: Paper-based data collection
- Web-based data collection (Active Comparator): Web-based data collection
  Interventions: Other: Web-based data collection

INTERVENTIONS:
Other: Web-based data collection
  Arms: Web-based data collection
Other: Paper-based data collection
  Arms: Paper-based data collection

SUMMARY:
This is an observational study to determine the effect of various treatments prescribed by healthcare providers for heavy menstrual bleeding on bleeding related quality of life (as measured by the Menstrual Bleeding Questionnaire) and to compare electronic and paper-based modes of data collection.

DETAILED DESCRIPTION:
Approximately 10% of women of reproductive age seek medical care each year for evaluation and treatment of heavy menstrual bleeding. Women with heavy menstrual bleeding suffer diminished quality of life, [1-2] lose work productivity,[3] and utilize expensive medical resources.[4] Although hysterectomy is considered the "definitive" treatment for heavy menstrual bleeding, many other options are available including endometrial ablation, the levonorgestrel intrauterine system (LNG-IUS), combined oral contraceptives (COCs), oral progestin, NSAIDs, and tranexamic acid. Better characterization of the relative efficacy of commonly used therapies for abnormal uterine bleeding will improve patient counseling, facilitate informed decision-making, and reduce the burden of unnecessary procedures on both the patient and the health care system. The data comparing these treatments in terms of patient-based outcome measures and bleeding-related quality of life are quite limited. We plan to prospectively compare bleeding-related quality of life between treatment methods within a cohort of patients receiving clinical care for heavy menstrual bleeding.

This study is being performed to determine the effect of various treatments prescribed by healthcare providers for heavy menstrual bleeding on bleeding related quality of life (as measured by the MBQ) and to compare electronic and paper-based modes of data collection. Eligible and consenting participants will be randomized to complete the study questionnaires electronically on IPad devices or on paper. At enrollment, participants will complete a background questionnaire and the MBQ. The background questionnaire will include information on age, race-ethnicity, primary language, income, education, and other medical issues. (Background Information Form) This will allow us to evaluate the effect of important demographic characteristics and concomitant medical problems on the effectiveness of prescribed treatments for heavy menstrual bleeding. We will also perform a chart review to validate the patient-reported medical information.

This study includes both prospective data collection with randomization of participants to mode of data collection. Studies will be conducted at Women and Infants Hospital in the Women's Primary Care Center. Approximately 13,000 women are seen for care that is not related to pregnancy. If only 10% of these women report heavy menstrual bleeding (which has a prevalence of 10-30%), 1300 patients in the WPCC could be eligible for these studies annually. Patient charts will be reviewed for potential eligibility in the WPCC in the evening and the morning. We plan to approach patients for screening who are presenting for gynecologic visits or well-woman examinations who still have an intact uterus and are between the ages of 18 and 51 years. The research assistant will make a list of names and appointment times to plan recruitment and will place a note on the front of the chart to page her when the patient is placed in a room. Lists of names will be destroyed each day. The research assistant or principal investigator will approach patients and screen them for eligibility. (Screening Form) The study will be described to eligible participants and informed consent obtained.

ELIGIBILITY:
Inclusion Criteria:

Patients who are presenting for gynecologic visits or well-woman examinations who still have an intact uterus and are between the ages of 18 and 51 years, have abnormal uterine bleeding, and can read and write in English.

Exclusion Criteria:

* Women who are presently on a treatment for abnormal uterine bleeding.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2015-07 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Menstrual bleeding questionnaire score | 6 months
  Condition-specific quality of life measurement tool for heavy menstrual bleeding compare change in quality of life over time between women receiving different treatments for heavy menstrual bleeding

SECONDARY OUTCOMES:
Quality of data collected | 6 Months
  Compare between the two modes of data collection(paper and electronic):
  number of "unusable" answers correlation of item responses to domain scores

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Matteson, MD, MPH, Principal Investigator — Women & Infants Hospital, Brown University
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States